CLINICAL TRIAL: NCT07082062
Title: Exploring the Effects of GLP-1 Formula on GLP-1 Secretion and Postprandial Glucose Regulation
Brief Title: Effects of GLP-1 Formula on GLP-1 and Glucose Regulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shih Chien Huang (Other)
Collaborators: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Shih Chien Huang, PhD, Assistant Professor, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CS2-24173
Record Dates: First submitted 2025-06-30; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Overweight
Keywords: Probiotic; Prebiotic; Glucagon-like peptide-1 (GLP-1); Blood glucose; Insulin
MeSH Terms: conditions — Overweight; Insulin Resistance | interventions — Arabinose; Erythritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Participants in the control group will consume 100 mL water
- GLP-1 formula Group (Experimental): Participants in the intervention group will consume a single dose of GLP-1 formula drink (50 mL) on the study day. The formula includes Bifidobacterium breve (probiotic), ClpB formula (prebiotic), and Rocket Apple extract.
  Interventions: Dietary Supplement: GLP-1 formula Group

INTERVENTIONS:
Dietary Supplement: GLP-1 formula Group — Participants in the intervention group will consume a single dose of GLP-1 formula drink (50 mL) on the study day. The formula includes Bifidobacterium breve (probiotic), ClpB formula (prebiotic), and Rocket Apple extract. The ClpB formula consists of kombucha, soy peptide powder, L-arabinose and erythritol.
  Other Names: Bifidobacterium breve; ClpB formula consists of kombucha, soy peptide powder, L-arabinose and erythritol.; Rocket Apple extract
  Arms: GLP-1 formula Group

SUMMARY:
This clinical trial is designed to evaluate the physiological effects of a GLP-1 Formula on glucagon-like peptide-1 (GLP-1) secretion and glycemic regulation in adults with elevated body fat percentage. The GLP-1 Formula is a multi-component dietary supplement composed of Bifidobacterium breve (probiotic), ClpB Formula-a prebiotic blend containing probiotic kombucha extract, soy peptide powder, L-arabinose, and erythritol-and rocket apple extract. The study consists of two randomized crossover trials: Trial 1 (n = 50) aims to assess the effects of the formula on circulating GLP-1 concentrations, while Trial 2 (n = 50) investigates its impact on blood glucose and insulin responses.

Eligible participants will be healthy adults aged 18 to 50 years with a body fat percentage greater than 25%, recruited via institutional and online outreach. Participants may choose to enroll in either or both trials; if enrolled in both, a washout period of at least one month between trials is required. Each trial consists of two intervention visits following a crossover design, with supplementation switched on day 8. Each visit will last approximately 6 hours, during which physiological and biochemical assessments will be conducted. Primary outcome measures include plasma levels of GLP-1, glucose, and insulin; secondary outcomes include appetite-related indices. This study aims to elucidate the potential of this functional formula to modulate incretin response and glycemic homeostasis in individuals with elevated adiposity.

DETAILED DESCRIPTION:
This study investigates the physiological effects of a multi-component GLP-1 Formula on incretin secretion and glycemic regulation in overweight adults. GLP-1, a key incretin hormone, plays a critical role in enhancing insulin secretion, suppressing glucagon release, and reducing appetite, making it a promising target in metabolic health modulation. The GLP-1 Formula under investigation includes Bifidobacterium breve (a probiotic strain), ClpB Formula (a prebiotic mixture composed of kombucha extract, soy peptide powder, L-arabinose, and erythritol), and rocket apple extract, which together are hypothesized to act synergistically to promote endogenous GLP-1 secretion and improve postprandial glucose control.

The study consists of two randomized crossover trials. Trial 1 aims to evaluate the acute effects of the formula on plasma GLP-1 concentrations following a single oral dose. Trial 2 investigates the impact of the formula on postprandial glucose and insulin responses under similar controlled conditions. Participants will undergo two intervention visits in each trial, with a washout period between them. Each visit will last approximately six hours, during which fasting and postprandial blood samples will be collected. In addition to biochemical endpoints, appetite-related indices will also be assessed to explore the formula's potential effect on satiety.

This investigation aims to provide foundational clinical evidence regarding the efficacy of functional dietary components in modulating incretin response and glycemic homeostasis, which may inform future development of non-pharmacological strategies for metabolic regulation in populations with elevated adiposity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18-50 years with a body fat percentage greater than 25%.

Exclusion Criteria:

* Use of probiotics, weight loss products, or gastrointestinal health-related supplements or medications within the past month.
* Presence of diabetes, autoimmune diseases, cancer, chronic gastrointestinal disorders, lactose intolerance, or chronic diarrhea.
* History of gastrointestinal surgery.
* Pregnant or breastfeeding women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma GLP-1 concentration (pmol/L) | Day 1 and Day 7
  Plasma GLP-1 levels will be measured at fasting and at 15, 30, 45, 60, 90, 120, and 240 minutes after consumption of the GLP-1 Formula on Days 1 and 7.
Blood glucose concentration (mg/dL) | Day 1 and Day 7
  Blood glucose levels will be measured at fasting and at 15, 30, 45, 60, 90, 120, and 240 minutes after consumption of the GLP-1 Formula on Days 1 and 7.
Serum insulin concentration (μIU/mL) | Day 1 and Day 7
  Serum insulin levels will be measured at fasting and at 15, 30, 45, 60, 90, 120, and 240 minutes after consumption of the GLP-1 Formula on Days 1 and 7.

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Chien Huang, PhD, Associate Professor, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD)